CLINICAL TRIAL: NCT03505931
Title: Korean Multicenter Registry of ELUVIA Stent for Femoropopliteal Artery Disease (K-ELUVIA Registry)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2015-0095
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Symptomatic Peripheral Artery Disease With Femoropopliteal Lesions; Moderate or Severe Claudication (Rutherford Category 2 or 3); Critical Limb Ischemia (Rutherford Category 4 or 5)
Keywords: Peripheral artery disease; femoropopliteal; drug-eluting stent; restenosis
MeSH Terms: conditions — Lymphoma, Follicular; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eluvia: Patients treated with Eluvia stent
  Interventions: Device: Implantation of Eluvia stent

INTERVENTIONS:
Device: Implantation of Eluvia stent — Implantation of Eluvia stent

SUMMARY:
* Prospective, multi-center single-arm observational study
* A total of 100 subjects with femoropopliteal artery disease who meet all inclusion and exclusion criteria will be included.
* Patients will be followed clinically for 12 months after the procedure.
* An imaging study (duplex ultrasound, CT or catheter-based angiography) follow-up according to participating hospital's protocol will be performed at 12 months.
* Ankle-brachial index, symptom status and presence of stent fracture will be evaluated at 12 months.

DETAILED DESCRIPTION:
Enrollment (day 0):

1) Written consent

Post PTA (Day 1 ~3):

1. Symptom: Rutherford class
2. Adverse event
3. Ankle-brachial index
4. Laboratory test: - eGFR, Cr, ALT, AST

   * Hb, WBC, platelet
5. Concomitant medication

Regular Follow-up Visits

Visit 1 (post-PTA 30±14 days):

1. Symptom: Rutherford class
2. Physical examination
3. Concomitant medication
4. Adverse event
5. Laboratory test:

   * AC glucose, eGFR, Cr, ALT, AST
   * Hb, WBC, platelet
   * Lipid level (total cholesterol, LDL-C, triglyceride, HDL-C)
   * HbA1c in case of DM
   * hsCRP

Visit 2 (post-PTA 6 months ± 30 days):

1. Symptoms: Rutherford class
2. Physical examination
3. Ankle-brachial index
4. Concomitant medication
5. Adverse event

Visit 3 (post-PTA 12 months ± 30 days): (Mandatory)

1. Symptoms: Rutherford class
2. Physical examination
3. Ankle-brachial index
4. Duplex ultrasound, CT, or catheter angiography
5. Concomitant medication
6. Adverse event 7) Biplane radiograph of femur for evaluation of stent fracture 8) Laboratory test: - AC glucose, eGFR, Cr, ALT, AST

   * Hb, WBC, platelet
   * Lipid level (total cholesterol, LDL-C,triglyceride, HDL-C)
   * HbA1c in case of DM
   * hsCRP

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years of older
* Symptomatic peripheral artery disease: Moderate or severe claudication (Rutherford category 2 or 3) and Critical limb ischemia (Rutherford category 4-5)
* Femoropopliteal artery lesions with stenosis > 50%
* ABI < 0.9 before treatment
* Patents treated with ELUVIA stent for femoropopliteal artery disease
* Patients with signed informed consent

Exclusion Criteria:

* Acute critical limb ischemia
* Severe critical limb ischemia (Rutherford category 6)
* Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, cilostazol, or contrast agents
* In-stent restenosis lesions (Restenosis lesions without previously implanted stents are eligible to the enrollment)
* Bypass graft lesions
* Age > 85 years
* Severe hepatic dysfunction (> 3 times normal reference values)
* Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* LVEF < 40% or clinically overt congestive heart failure
* Pregnant women or women with potential childbearing
* Life expectancy <1 year due to comorbidity
* Untreated proximal inflow disease of the ipsilateral iliac arteries (more than 50% stenosis or occlusion)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic peripheral artery disease with femoropopliteal lesions:
  * Moderate or severe claudication (Rutherford category 2 or 3)
  * Critical limb ischemia (Rutherford category 4 or 5) Age: ≥19 years, but not older than 85 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Primary patency | at 12 months
  Absence of stenosis >50% by an follow-up imaging study (duplex ultrasound, CT or catheter-based angiography) at 12 months

SECONDARY OUTCOMES:
Ankle-brachial index | at 12 months
  Ankle-brachial index defined as the ratio of the blood pressure at the ankle to the blood pressure in the upper arm
Ruthford category | at 12 months
  Rutherford category - symptom status by Rutherford category
target lesion revascularization | at 12 months
  Target lesion revascularization - accumulative rate of repeat interventions or surgery for the treatment of symptomatic restenosis (>50% stenosis) in the target lesion
stent fracture rate | at 12 months
  stent fracture rate - incidence of stent fracture by radiographs or fluoroscopy in 2 different projections

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided